CLINICAL TRIAL: NCT03729492
Title: Symptom-driven Referral for Evaluation of Chronic Thromboembolic Disease or Pulmonary Hypertension in Patients With Previous Acute Pulmonary Embolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Hospitalsenheden Vest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTEPH
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Chronic Thromboembolic Pulmonary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTEPH/CTED work-up (Other)
  Interventions: Diagnostic Test: CTEPH/CTED work-up

INTERVENTIONS:
Diagnostic Test: CTEPH/CTED work-up — Patients diagnosed with acute pulmonary embolism (PE) in Region Midt (approx. 350 per year) will be screened for non-recovery or persistent PE related symptoms during their 3-6 months follow up at their local outpatient clinic. If the patient has persistent symptoms they will be referred to a V/Q-scan. If a V/Q mismatch is present, the patient will be referred to a full work-up for CTEPH/CTED.

SUMMARY:
Aim: To investigate if a symptom driven referral for chronic thrombosis in the lungs after acute pulmonary embolism is better than the current approach.

Background: A number of patients with chronic thrombosis in the lungs after acute pulmonary embolism have dyspnea and reduced functional capacity without elevated pulmonary arterial pressure at rest (CTED). However, current guidelines for follow-up after acute pulmonary embolism will miss all patients with CTED, as referral for further examination is based on elevated pulmonary arterial pressure on echocardiography. Thus, the prevalence of CTED is unknown. The hypothesis is, that a symptom-driven referral of patients with previous acute pulmonary embolism is more sensitive in diagnosing CTED than the current approach.

Methods and materials: Patients diagnosed with acute pulmonary embolism in Region Midt (approx. 350 per year) will be screened for non-recovery or persistent pulmonary embolism related symptoms during their 3-6 months follow up at their local outpatient clinic. If the patient has persistent symptoms they will be referred to a scintigraphy. If CTED is suspected from the scintigraphy, the patient will be referred for full CTED work-up. The investigators expect to screen 300 patients for persistent symptoms with an expected study time of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute PE diagnosed by CT or V/Q-scan within the last year.
* Non-recovery or persistent PE related symptoms assessed by a MRC breathlessness score or WHO functional class.
* Age >= 18 and < 80

Exclusion Criteria:

* Contraindications or unable to perform 6 minutes walk distance (6MWD) and/or cardiopulmonary exercise test.
* Contraindications to CT pulmonary angiography.
* Congestive heart failure (LVEF <40%).
* COPD or restrictive lung disease, severe or worse (FEV1 <50% and >=1 exacerbation causing hospital admission per year (GOLD grade 3 and 4 class C and D)).
* Lactating or pregnant.
* Unable or unwilling to provide written informed consent.
* Paroxysmal or persistent atrial fibrillation.
* Other known cause of PE related symptoms.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CTED | 3 years

SECONDARY OUTCOMES:
Diagnostic accuracy of dual energy CT perfusion and pulmonary angiography. | 3 years
  Sensibility, specificity, positive predictive value and negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Asger Andersen, MD, PhD, Study Chair — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: No